CLINICAL TRIAL: NCT00715156
Title: Classification of Different Forms of Peach Allergy and the Role of Recombinant Allergens in the Diagnosis
Brief Title: Role of Recombinants in Peach Allergy
Status: Completed | Type: Observational
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Peach allergy
Record Dates: First submitted 2008-07-14; First posted 2008-07-15 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Food Allergy
Keywords: allergy, peach, birch; recombinants allergens diagnosis; OAS; LTP; systemic reactions; subjects with severe reaction to other fruits
MeSH Terms: conditions — Food Hypersensitivity; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: Subjects with mild (S1) reaction to peach fruit
- B: Subjects with severe reaction to peach fruit

SUMMARY:
This study is aimed at verifying the role and the efficacy of the recombinants allergens Pru p 1, Pru p 3 and Pru p 4, Bet v 1, Bet v 2 and Bet v 4 in the diagnosis of peach allergy

DETAILED DESCRIPTION:
This study intend to verify whether the different levels of severity of the clinical allergic reactions to peach are associated to sensitization towards different allergenic molecules of peach. In particular, we will analyze the reactivity towards the peach allergens Pru p 1, Pru p 3 and Pru p 4 and towards the birch pollen allergens Bet v 1, Bet v 2 and Bet v 4. The patients (with allergic symptoms of any severity provoked by the consumption of peach) will be divided into two groups: the first group showing oral allergy syndrome (OAS), the second group showing systemic symptoms of different severity, up to anaphylaxis.

All the patients will be submitted to: complete clinical investigation; skin prick test with a panel of common food/inhalant commercial extracts; skin tests by the "prick + prick" method with fresh fruits and vegetables; skin prick test with purified peach LTP (Pru p 3) The sera of the patients will be used for: immunoblotting with peach extract and immunoblotting inhibition with purified natural Pru p 3 and, if possible, recombinant Pru p 3, Pru p 1 and Pru p 4, using a pool of selected sera; CAP system with a predetermined panel of fruit and vegetable allergens; CAP system with recombinant allergens of peach and birch pollen: Pru p 3, Pru p 1 and Pru p 4 for peach, Bet v 1, Bet v 2 and Bet v 4 for birch pollen. Finally, a statistical analysis will be carried out in order to verify if the two groups of patients will show significant differences in the allergens recognized. The results of this study will be a property of the Unit of Allergology and Immunology as stated by DM 17/2004 and will be presented as written publication or oral presentation at National and/or International Congresses of Allergy and Immunology, quoting the PHADIA company

ELIGIBILITY:
Inclusion Criteria:

* female and male;
* pts with 18 e 80 years old;
* signature of the informed consent form;
* CAP/RAST positive for peach;
* clinical manifestation of peach allergy

Exclusion Criteria:

* pregnancy;
* current antihistamine therapy;
* subjects that do not give consent to the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Peach allergic subjects at major risk of anaphylaxis
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2008-07; Primary Completion 2009-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of diagnostic efficacy of PHADIA IMMUNO-CAP with the peach recombinant allergens Pru p 3, 1 and 4 as compared to peach IMMUNO-CAP in the identification of peach allergic subjects at major risk of anaphylaxis | 1 year

SECONDARY OUTCOMES:
Evaluate whether the above recombinants allergens could help identifying subjects with severe reaction to other fruits | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Elide A Patorello, MD, Principal Investigator — Niguarda Hospital
Locations (1):
- Niguarda Hospital, Milan, Italy, Italy

REFERENCES:
- [Result] Pastorello EA, Farioli L, Pravettoni V, Scibilia J, Mascheri A, Borgonovo L, Piantanida M, Primavesi L, Stafylaraki C, Pasqualetti S, Schroeder J, Nichelatti M, Marocchi A. Pru p 3-sensitised Italian peach-allergic patients are less likely to develop severe symptoms when also presenting IgE antibodies to Pru p 1 and Pru p 4. Int Arch Allergy Immunol. 2011;156(4):362-72. doi: 10.1159/000324440. Epub 2011 Aug 9. PMID 21829031
- [Derived] Mascheri A, Farioli L, Pravettoni V, Piantanida M, Stafylaraki C, Scibilia J, Mirone C, Preziosi D, Nichelatti M, Pastorello EA. Hypersensitivity to Tomato (Lycopersicon esculentum) in Peach-Allergic Patients: rPrup 3 and rPrup 1 Are Predictive of Symptom Severity. J Investig Allergol Clin Immunol. 2015;25(3):183-9. PMID 26182684